CLINICAL TRIAL: NCT06117735
Title: A Prospective, Multicenter, Single-arm Clinical Study of PTFE Covered Stent for Treating Portal Hypertension.
Brief Title: Clinical Study of PTFE Covered Stent for Treating Portal Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enlight Medical Technologies (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YM-2023-002
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Portal Hypertension
Keywords: transjugular intrahepatic portosystemic shunt
MeSH Terms: conditions — Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTFE covered stent (Experimental): Use the experimental device, PTFE covered stent to treat protal hypertension.
  Interventions: Device: Transjugular Intrahepatic Portosystemic shunt

INTERVENTIONS:
Device: Transjugular Intrahepatic Portosystemic shunt — The experimental device is a class III implanted shunt device, which will be used to create a shunt between intrahepatic and portosystemic to reduce portal hypertension.

SUMMARY:
To validate the safety and efficacy of TIPS (Transjugular Intrahepatic Portosystemic Shunt) using PTFE covered stent in the treatment of portal hypertension.

DETAILED DESCRIPTION:
This trial is a prospective multi-center single-arm confirmatory study. A total 177 subjects will be enrolled in multiple centers nationwide. Subjects who meet the trial requirements, fulfill the inclusion criteria, voluntarily participate in the study, and provide informed consent will undergo TIPS using the PTFE covered stent for the treatment of portal hypertension. Follow-up assessments will be conducted at discharge, as well as at 30 days, 90 days, 180 days and 360 days postoperatively. Secondary endpoint measures include surgical success rate, all-cause mortality, device/procedure-related mortality, incidence of adverce events, and serious adverse event rates. The trial aims to comprehensively assess the safety and efficacy of the PTFE covered stent produced by Enlight Medical Technologies (Shanghai) Co., Ltd..

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for this study:

* Age 18-85 years;
* Cirrhotic portal hypertension required for TIPS;
* Willingness to comply with the protocol requirements and ata collection procedures, ability to understand the purpose of the trial, voluntary participation, and signing of informed consent by the subject or legal guardian.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for this study:

* Concomitant chronic heart or lung disease;
* Presence or suspicion of active systemic, hepatobiliary or ascitic fluid infection;
* Severe hepatic failure (with bilirubin levels of >51.3μmol/L or Child-Pugh >13 or MELD >18);
* Hepatic encephalopathy;
* Coagulation disorders;
* Portal vein thrombosis;
* Allergies to device components;
* Extrahepatic malignancy;
* Pregnant or brestfeeding women or those planning pregnancy during the trial peroid;
* Intending or currently participating in another interventional clinical trial;
* Other conditions deemed inappropriate for participation in this study by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary shunt patency rate | 1 year
  shunt dysfunction was defined as a TIPS stenosis >=50% or complete occlusion. Primary patency referred to continuous unassisted patency of the shunt.

SECONDARY OUTCOMES:
Technical success rate | immediately after procedure
  Successful implantation of a PTFE covered stent to create an intrahepatic portosystemic shunt and successful retrieval of the delivery system.
Procedure success rate | immediately after procedure
  PPG (portosystemic pressure gradient) reduces more than 20% or PPG <=12mmHg
Treatment success rate | during the perioperative period
  Treatment success is defined as the success of the procedure without major adverse event.

OTHER OUTCOMES:
Secondary patency rate | 1 year
  Second patency was defined as graft stenosis or occlusion with patency restored and maintained by TIPS revision.
all cause mortalidy | through study completion, an average of 1 year
Device-related adverse events | through study completion, an average of 1 year
Serious adver events | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bin Xiong, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (4):
- China (4):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The first affiliated hospital of Guangzhou Medical University, Guangzhou, Guangzhou
  - Shanghai Public Health Clinical Center, Shanghai, Jinshan
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi